CLINICAL TRIAL: NCT04437407
Title: UniSA BackOff! Study: A Randomized, Controlled, Five-way, Cross-over Trial to Evaluate the Effect of a Positional Therapy Device on Maternal Sleeping Position in the Third Trimester of Pregnancy
Brief Title: UniSA BackOff! Study: Adelaide PrenaBelt Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant dropout and technical difficulties
Sponsor: Shiphrah Biomedical Inc. (Industry)
Collaborators: University of South Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 202902
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Stillbirth; Infant, Low Birth Weight; Infant, Very Low Birth Weight; Sleep-Disordered Breathing; Infant, Small for Gestational Age; Fetal Hypoxia; Pregnancy Complications; Fetal Growth Retardation
Keywords: Pregnancy; Sleep; Maternal
MeSH Terms: conditions — Stillbirth; Sleep Apnea Syndromes; Fetal Hypoxia; Pregnancy Complications; Fetal Growth Retardation

STUDY DESIGN:
Intervention Model Description: A consecutive, six-night, in-home, controlled, cross-over sleep study in third-trimester pregnant women to validate the ability of the PB2 and Ajuvia devices to reduce the amount of time pregnant women spend sleeping on their backs at night in the home setting in the third trimester of pregnancy
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (Other): The first night will be a control night with infrared video recording where only the Ajuvia sleep monitor is worn in passive mode so that each participant can act as her own control for comparison of treatment effect on outcomes.
  Interventions: Device: Ajuvia-Passive
- PB2-1 (Experimental): During this night, the PB2-1 prototype will be worn with the Ajuvia in passive mode.
  Interventions: Device: PB2-1 prototype; Device: Ajuvia-Passive
- PB2-2 (Experimental): During this night, the PB2-2 prototype will be worn with the Ajuvia in passive mode.
  Interventions: Device: PB2-2 prototype; Device: Ajuvia-Passive
- PB2-3 (Experimental): During this night, the PB2-3 prototype will be worn with the Ajuvia in passive mode.
  Interventions: Device: PB2-3 prototype; Device: Ajuvia-Passive
- PB2-4 (Experimental): During this night, the PB2-4 prototype will be worn with the Ajuvia in passive mode.
  Interventions: Device: PB2-4 prototype; Device: Ajuvia-Passive
- PB2-5 (Experimental): During this night, the PB2-5 prototype will be worn with the Ajuvia in active mode.
  Interventions: Device: PB2-5 prototype; Device: Ajuvia-Active

INTERVENTIONS:
Device: PB2-1 prototype — PB2-1 prototype is a belt-like wearable device similar to the original PrenaBelt designed for pregnant women that permits supine positioning of the pelvis but, when in this position, provides subtle pressure points to the user's body and thereby activates the body's natural mechanism to reposition itself to relieve discomfort. It is expected to significantly decrease the amount of time a pregnant woman's pelvis is in the supine position overnight while promoting comfortable sleep.
  Arms: PB2-1
Device: PB2-2 prototype — PB2-2 prototype is a belt-like wearable device designed for pregnant women. When placed on the woman's back, this device prevents the pelvis from achieving a supine orientation by maintaining at least fifteen degrees of right or left lateral pelvic tilt. It is expected to significantly decrease the amount of time a pregnant woman's pelvis is in the supine position overnight while promoting comfortable sleep.
  Arms: PB2-2
Device: PB2-3 prototype — PB2-3 prototype is a belt-like wearable device designed for pregnant women. When placed on the woman's back, this device prevents the pelvis from achieving a supine orientation by maintaining at least fifteen degrees of right or left lateral pelvic tilt. It is expected to significantly decrease the amount of time a pregnant woman's pelvis is in the supine position overnight while promoting comfortable sleep.
  Arms: PB2-3
Device: PB2-4 prototype — PB2-4 prototype is a belt-like wearable device designed for pregnant women that prevents the user from achieving a supine position as the device allows right and left lateral pelvic tilt but prevents the user's pelvis from settling supine due to virtue of its design. It is expected to significantly decrease the amount of time a pregnant woman's pelvis is in the supine position overnight while promoting comfortable sleep.
  Arms: PB2-4
Device: PB2-5 prototype — PB2-5 prototype is a belt-like wearable device designed for pregnant women that does not provide positional therapy. It can be worn anytime as a maternity support belt.
  Arms: PB2-5
Device: Ajuvia-Active — Ajuvia Sleep Monitor senses the user's body position and can be used in passive or active mode with or without the PB2 prototypes. In the active mode, it alerts the woman when her pelvis is in the supine position through a gentle vibratory alarm.
  Arms: PB2-5
Device: Ajuvia-Passive — Ajuvia Sleep Monitor senses the user's body position and can be used in passive or active mode with or without the PB2 prototypes. In the passive mode, it measures and records the position of the pelvis but does not alert the woman.
  Arms: Control; PB2-1; PB2-2; PB2-3; PB2-4

SUMMARY:
Stillbirth (SB) is a devastating complication of pregnancy and contributes to over 2 million deaths globally every year. Over 20 million infants are born every year with low birth weight (LBW), which is associated with a twenty times increased risk of death in the first year of life and high rates of short- and long-term illnesses. Sleeping on one's back during pregnancy has recently emerged as a potential risk factor for LBW and SB in the medical literature. In high-income countries, SB rates have mostly remained the same in the past two decades and targeting modifiable risk factors could help reduce the number of SB and LBW in the population.

When a pregnant woman sleeps on her back, her body position compresses underlying blood vessels and reduces blood flow to the developing baby. This body position could cause unpleasant symptoms for the mother and result in LBW or SB of her baby. Lying on her side or with a slight lateral tilt helps relieve this compression. One way to keep people off their back while sleeping is by using positional therapy (PT). It is a simple, safe, inexpensive and effective intervention for preventing people who snore or people who's breathing pauses during sleep from sleeping on their back. Reducing the amount of time pregnant women sleep on their back could help reduce SB and LBW rates. The investigators developed a PT device (PrenaBelt) and tested it in three clinical trials, which demonstrated that it significantly decreases the number of time women spend sleeping on their back. Using feedback from our previous research, the investigators developed five additional devices that will be tested in this study.

The purpose of this study is to evaluate the new PrenaBelt (PB2) prototypes' ability to reduce the amount of time pregnant women sleep on their backs in the third trimester of pregnancy, validate the Ajuvia Sleep Monitor, and collect feedback on the devices.

Demonstrating that the sleeping position of pregnant women can be modified through the use of a simple, inexpensive PT intervention may be one of the keys to achieving significant reductions in LBW and late SB rates in Australia and worldwide.

DETAILED DESCRIPTION:
The ability of the PB2 prototypes to reduce the amount of time pregnant women spend sleeping on their backs at night in the home setting in the third trimester of pregnancy will be evaluated via a consecutive, six-night, in-home, controlled, cross-over sleep study in third trimester pregnant women where the Ajuvia Sleep Monitor is validated against infrared video on the first night.

Six nights: the first night is a control night with infrared video recording where only the Ajuvia is worn in passive mode to collect data on the participant's body position and is followed by five nights with the five different prototypes.

Randomization: The order in which the different devices will be worn on the second night through fourth night, inclusive, will be determined by simple randomization. This will minimize the potential impact of changes to sleep across the nights resulting from familiarization with the equipment as the sleep tests proceed through the five non-control nights, which could bias the results. For logistical reasons, the sixth night is non-randomized and will include the Ajuvia in 'active' mode Cross-over: After the first night, on each of the subsequent four nights, the participants will "cross over" to a different PB2 device (depending on their randomization order) and "cross over" to the Ajuvia in 'active' mode on the sixth night to allow each participant to act as her own control for comparison of treatment effect on outcomes.

In home: conducting this study in the home setting will allow for a more accurate representation of sleep patterns as the participants will be in the comfort of their own bed.

Sleep test: The maternal pelvis position will be recorded while the participants are sleeping using the Ajuvia device. Going to bed- and wake-times, as well as experience with each device will be recorded daily in a sleep diary.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* low-risk singleton pregnancy
* in the last trimester of pregnancy (at least 28 weeks + 0 days but not more than 36 weeks + 0 days of gestation)
* access to and ability to use iPhone (for downloading and using Ajuvia app)
* residing in the Greater Adelaide Area.

Exclusion Criteria:

* musculoskeletal disorder that prevents sleeping supine or on a certain side (e.g., arthritic shoulder)
* non-English speaking and reading

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Ajuvia for supine position | 1 night (approximately 8 hours)
  The sensitivity(%) of the Ajuvia in determining the pelvic supine position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Specificity of Ajuvia for supine position | 1 night (approximately 8 hours)
  The specificity(%) of the Ajuvia in determining the pelvic supine position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Sensitivity of Ajuvia for prone position | 1 night (approximately 8 hours)
  The sensitivity(%) of the Ajuvia in determining the pelvic prone position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Specificity of Ajuvia for prone position | 1 night (approximately 8 hours)
  The specificity(%) of the Ajuvia in determining the pelvic prone position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Sensitivity of Ajuvia for left tilt position | 1 night (approximately 8 hours)
  The sensitivity(%) of the Ajuvia in determining the left pelvic tilt position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Specificity of Ajuvia for left tilt position | 1 night (approximately 8 hours)
  The specificity(%) of the Ajuvia in determining the left pelvic tilt position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Sensitivity of Ajuvia for left lateral position | 1 night (approximately 8 hours)
  The sensitivity(%) of the Ajuvia in determining the left lateral pelvic position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Specificity of Ajuvia for left lateral position | 1 night (approximately 8 hours)
  The specificity(%) of the Ajuvia in determining the left lateral pelvic position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Sensitivity of Ajuvia for right tilt position | 1 night (approximately 8 hours)
  The sensitivity(%) of the Ajuvia in determining the right pelvic tilt position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Specificity of Ajuvia for right tilt position | 1 night (approximately 8 hours)
  The specificity(%) of the Ajuvia in determining the right pelvic tilt position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Sensitivity of Ajuvia for right lateral position | 1 night (approximately 8 hours)
  The sensitivity(%) of the Ajuvia in determining the right lateral pelvic position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Specificity of Ajuvia for right lateral position | 1 night (approximately 8 hours)
  The specificity(%) of the Ajuvia in determining the right lateral pelvic position during night sleep against the gold-standard of position as determined by review of infrared video will be calculated using a two-by-two contingency table.
Supine Sleep Time - Control | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the supine position with Ajuvia in passive mode
Supine Sleep Time - PB2-1 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the supine position with PB2-1 and Ajuvia in passive mode
Supine Sleep Time - PB2-2 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the supine position with PB2-2 and Ajuvia in passive mode
Supine Sleep Time - PB2-3 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the supine position with PB2-3 and Ajuvia in passive mode
Supine Sleep Time - PB2-4 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the supine position with PB2-4 and Ajuvia in passive mode
Supine Sleep Time - PB2-5 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the supine position with PB2-5 and Ajuvia in active mode
Prone Sleep Time - Control | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the prone position with Ajuvia in passive mode
Prone Sleep Time - PB2-1 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the prone position with PB2-1 and Ajuvia in passive mode
Prone Sleep Time - PB2-2 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the prone position with PB2-2 and Ajuvia in passive mode
Prone Sleep Time - PB2-3 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the prone position with PB2-3 and Ajuvia in passive mode
Prone Sleep Time - PB2-4 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the prone position with PB2-4 and Ajuvia in passive mode
Prone Sleep Time - PB2-5 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the prone position with PB2-5 and Ajuvia in active mode
Left-tilt Sleep Time - Control | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left pelvic tilt position with Ajuvia in passive mode
Left-tilt Sleep Time - PB2-1 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left pelvic tilt position with PB2-1 and Ajuvia in passive mode
Left-tilt Sleep Time - PB2-2 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left pelvic tilt position with PB2-2 and Ajuvia in passive mode
Left-tilt Sleep Time - PB2-3 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left pelvic tilt position with PB2-3 and Ajuvia in passive mode
Left-tilt Sleep Time - PB2-4 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left pelvic tilt position with PB2-4 and Ajuvia in passive mode
Left-tilt Sleep Time - PB2-5 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left pelvic tilt position with PB2-5 and Ajuvia in active mode
Left-lateral Sleep Time - Control | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left lateral position with Ajuvia in passive mode
Left-lateral Sleep Time - PB2-1 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left lateral position with PB2-1 and Ajuvia in passive mode
Left-lateral Sleep Time - PB2-2 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left lateral position with PB2-2 and Ajuvia in passive mode
Left-lateral Sleep Time - PB2-3 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left lateral position with PB2-3 and Ajuvia in passive mode
Left-lateral Sleep Time - PB2-4 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left lateral position with PB2-4 and Ajuvia in passive mode
Left-lateral Sleep Time - PB2-5 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the left-lateral position with PB2-5 and Ajuvia in active mode
Right-tilt Sleep Time - Control | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right pelvic tilt position with Ajuvia in passive mode
Right-tilt Sleep Time - PB2-1 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right pelvic tilt position with PB2-1 and Ajuvia in passive mode
Right-tilt Sleep Time - PB2-2 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right pelvic tilt position with PB2-2 and Ajuvia in passive mode
Right-tilt Sleep Time - PB2-3 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right pelvic tilt position with PB2-3 and Ajuvia in passive mode
Right-tilt Sleep Time - PB2-4 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right pelvic tilt position with PB2-4 and Ajuvia in passive mode
Right-tilt Sleep Time - PB2-5 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right pelvic tilt position with PB2-5 and Ajuvia in active mode
Right-lateral Sleep Time - Control | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right lateral position with Ajuvia in passive mode
Right-lateral Sleep Time - PB2-1 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right lateral position with PB2-1 and Ajuvia in passive mode
Right-lateral Sleep Time - PB2-2 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right lateral position with PB2-2 and Ajuvia in passive mode
Right-lateral Sleep Time - PB2-3 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right lateral position with PB2-3 and Ajuvia in passive mode
Right-lateral Sleep Time - PB2-4 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right lateral position with PB2-4 and Ajuvia in passive mode
Right-lateral Sleep Time - PB2-5 | 1 night (approximately 8 hours)
  The time (in minutes) spent sleeping in the right lateral position with PB2-5 and Ajuvia in active mode

CONTACTS AND LOCATIONS:
Overall Officials: Jane Warland, PhD, Principal Investigator — University of South Australia
Locations (1):
- UniSA Clinical & Health Sciences, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kember AJ, Scott HM, O'Brien LM, Borazjani A, Butler MB, Wells JH, Isaac A, Chu K, Coleman J, Morrison DL. Modifying maternal sleep position in the third trimester of pregnancy with positional therapy: a randomised pilot trial. BMJ Open. 2018 Aug 29;8(8):e020256. doi: 10.1136/bmjopen-2017-020256. PMID 30158217
- [Background] Coleman J, Okere M, Seffah J, Kember A, O'Brien LM, Borazjani A, Butler M, Wells J, MacRitchie S, Isaac A, Chu K, Scott H. The Ghana PrenaBelt trial: a double-blind, sham-controlled, randomised clinical trial to evaluate the effect of maternal positional therapy during third-trimester sleep on birth weight. BMJ Open. 2019 May 1;9(4):e022981. doi: 10.1136/bmjopen-2018-022981. PMID 31048420
- [Background] Cronin RS, Li M, Thompson JMD, Gordon A, Raynes-Greenow CH, Heazell AEP, Stacey T, Culling VM, Bowring V, Anderson NH, O'Brien LM, Mitchell EA, Askie LM, McCowan LME. An Individual Participant Data Meta-analysis of Maternal Going-to-Sleep Position, Interactions with Fetal Vulnerability, and the Risk of Late Stillbirth. EClinicalMedicine. 2019 Apr 2;10:49-57. doi: 10.1016/j.eclinm.2019.03.014. eCollection 2019 Apr. PMID 31193832
- [Background] O'Brien LM, Warland J, Stacey T, Heazell AEP, Mitchell EA; STARS Consortium. Maternal sleep practices and stillbirth: Findings from an international case-control study. Birth. 2019 Jun;46(2):344-354. doi: 10.1111/birt.12416. Epub 2019 Jan 18. PMID 30656734
- [Background] Anderson NH, Gordon A, Li M, Cronin RS, Thompson JMD, Raynes-Greenow CH, Heazell AEP, Stacey T, Culling VM, Wilson J, Askie LM, Mitchell EA, McCowan LME. Association of Supine Going-to-Sleep Position in Late Pregnancy With Reduced Birth Weight: A Secondary Analysis of an Individual Participant Data Meta-analysis. JAMA Netw Open. 2019 Oct 2;2(10):e1912614. doi: 10.1001/jamanetworkopen.2019.12614. PMID 31577362
- [Background] Warland J, Dorrian J, Morrison JL, O'Brien LM. Maternal sleep during pregnancy and poor fetal outcomes: A scoping review of the literature with meta-analysis. Sleep Med Rev. 2018 Oct;41:197-219. doi: 10.1016/j.smrv.2018.03.004. Epub 2018 Mar 27. PMID 29910107
- [Background] Warland J, Dorrian J, Kember AJ, Phillips C, Borazjani A, Morrison JL, O'Brien LM. Modifying Maternal Sleep Position in Late Pregnancy Through Positional Therapy: A Feasibility Study. J Clin Sleep Med. 2018 Aug 15;14(8):1387-1397. doi: 10.5664/jcsm.7280. PMID 30092890
- [Background] McCowan LME, Thompson JMD, Cronin RS, Li M, Stacey T, Stone PR, Lawton BA, Ekeroma AJ, Mitchell EA. Going to sleep in the supine position is a modifiable risk factor for late pregnancy stillbirth; Findings from the New Zealand multicentre stillbirth case-control study. PLoS One. 2017 Jun 13;12(6):e0179396. doi: 10.1371/journal.pone.0179396. eCollection 2017. PMID 28609468
- [Background] Gordon A, Raynes-Greenow C, Bond D, Morris J, Rawlinson W, Jeffery H. Sleep position, fetal growth restriction, and late-pregnancy stillbirth: the Sydney stillbirth study. Obstet Gynecol. 2015 Feb;125(2):347-355. doi: 10.1097/AOG.0000000000000627. PMID 25568999
- [Background] Platts J, Mitchell EA, Stacey T, Martin BL, Roberts D, McCowan L, Heazell AE. The Midland and North of England Stillbirth Study (MiNESS). BMC Pregnancy Childbirth. 2014 May 21;14:171. doi: 10.1186/1471-2393-14-171. PMID 24885461
- [Background] Warland J, Mitchell EA. A triple risk model for unexplained late stillbirth. BMC Pregnancy Childbirth. 2014 Apr 14;14:142. doi: 10.1186/1471-2393-14-142. PMID 24731396
- [Background] O'Brien LM, Warland J. Typical sleep positions in pregnant women. Early Hum Dev. 2014 Jun;90(6):315-7. doi: 10.1016/j.earlhumdev.2014.03.001. Epub 2014 Mar 21. PMID 24661447
- [Background] Owusu JT, Anderson FJ, Coleman J, Oppong S, Seffah JD, Aikins A, O'Brien LM. Association of maternal sleep practices with pre-eclampsia, low birth weight, and stillbirth among Ghanaian women. Int J Gynaecol Obstet. 2013 Jun;121(3):261-5. doi: 10.1016/j.ijgo.2013.01.013. Epub 2013 Mar 15. PMID 23507553
- [Background] Stacey T, Thompson JM, Mitchell EA, Ekeroma AJ, Zuccollo JM, McCowan LM. Association between maternal sleep practices and risk of late stillbirth: a case-control study. BMJ. 2011 Jun 14;342:d3403. doi: 10.1136/bmj.d3403. PMID 21673002